CLINICAL TRIAL: NCT02775292
Title: NY-ESO-1 TCR Engineered Adoptive Cell Transfer Therapy With Nivolumab PD-1 Blockade
Brief Title: Gene-Modified T Cells, Vaccine Therapy, and Nivolumab in Treating Patients With Stage IV or Locally Advanced Solid Tumors Expressing NY-ESO-1
Acronym: NYM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Stand Up To Cancer (Other); Bristol-Myers Squibb (Industry); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-001433; NCI-2016-00201 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R35CA197633 (NIH); 15-001433 (Other: UCLA / Jonsson Comprehensive Cancer Center); K12HD000850 (NIH)
Record Dates: First submitted 2016-05-13; First posted 2016-05-17 (Estimated); Last update posted 2025-07-30 (Actual); Status verified 2019-08

CONDITIONS: Adult Solid Neoplasm; Childhood Solid Neoplasm; Metastatic Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — aldesleukin; Cyclophosphamide; fludarabine phosphate; Nivolumab; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (1):
- Treatment (NY-ESO-1 TCR transduced PBMC, vaccine, nivolumab) (Experimental): CONDITIONING REGIMEN: Patients receive cyclophosphamide IV over 1 hour on days -5 to -4 and fludarabine phosphate IV over 30 minutes on days -4 to -1.
  NY-ESO-1 TCR PBMC INFUSION: Patients receive NY-ESO-1 TCR PBMC IV on day 0.
  NIVOLUMAB: Patients receive nivolumab IV over 60 minutes on day 0 or 1. Treatment repeats every 2 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity.
  NY-ESO-1(157-165) PEPTIDE PULSED DC: Patients receive NY-ESO-1(157-165) peptide pulsed DC ID on days 1, 14, and 28.
  LOW DOSE ALDESLEUKIN ADMINISTRATION: Patients receive aldesleukin SC BID for 7 days beginning on day 1 for a maximum of 14 doses.
  Interventions: Biological: Aldesleukin; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Biological: Nivolumab; Biological: NY-ESO-1 Reactive TCR Retroviral Vector Transduced Autologous PBL; Biological: NY-ESO-1(157-165) Peptide-pulsed Autologous Dendritic Cell Vaccine; Procedure: Positron Emission Tomography

INTERVENTIONS:
Biological: Aldesleukin — Given SC
  Other Names: 125-L-Serine-2-133-interleukin 2; Proleukin; r-serHuIL-2; Recombinant Human IL-2; Recombinant Human Interleukin-2
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; Oforta; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Biological: NY-ESO-1 Reactive TCR Retroviral Vector Transduced Autologous PBL — Given IV
  Other Names: Anti-NY-ESO-1 TCR Retroviral Vector Transduced Autologous PBL
Biological: NY-ESO-1(157-165) Peptide-pulsed Autologous Dendritic Cell Vaccine — Given ID
  Other Names: Autologous NY-ESO-1 (157-165) Peptide-pulsed DC Vaccine
Procedure: Positron Emission Tomography — Correlative studies
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET SCAN; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This phase I trial studies the side effects and the best dose of nivolumab when given together with gene-modified T cells and vaccine therapy in treating patients with solid tumors that express the cancer-testes antigen NY-ESO-1 gene AND have spread from where it started to nearby tissue or lymph nodes (locally advanced) or distant organs (stage IV). T cells are a special type of white blood cells (immune cell) that have the ability to kill cancer cells. Nivolumab may block PD-1 which is found on T cells and help the immune system kill cancer cells. Placing a modified gene for the NY-ESO-1 T cell receptor (TCR) into the patients' T cells in the laboratory and then giving them back to the patient may help the body build an immune response to kill tumor cells that express NY-ESO-1. Dendritic cells are another type of blood cell that can teach other cells in the body to look for cancer cells and attack them. Giving a dendritic cell vaccine with the NY-ESO-1 protein may help dendritic cells teach the immune system to target cancer cells expressing that protein, and further help the T cells attack cancer. Giving nivolumab together with gene-modified T-cells and dendritic cell vaccine may teach the immune system to recognize and kill cancer cells that express NY-ESO-1.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety of the addition of the PD-1 blocking monoclonal antibody, nivolumab, to NY-ESO TCR-transduced autologous peripheral blood lymphocyte (PBL) adoptive cell transfer (ACT) in a dose escalation scheme in two study cohorts at 1 mg/kg and 3 mg/kg of nivolumab intravenous (i.v.) every two weeks for up to 2 years.

SECONDARY OBJECTIVES:

I. To determine the feasibility of delivering the TCR transgenic cell dose and PD-1 blockade to patients.

II. To determine the persistence of NY-ESO-1 TCR-engineered peripheral blood mononuclear cell (PBMC) in serial peripheral blood samples and in biopsies of accessible metastatic lesions.

EXPLORATORY OBJECTIVES:

I. To determine whether blocking PD-1 will maintain the antitumor functionality of adoptively transferred TCR transgenic lymphocytes.

II. To explore the use of positron emission tomography (PET)-based imaging using the PET tracer (18F) fluorodeoxy-glucose ([18F]FDG) with the goal of determining if the adoptively transferred NY-ESO-1 TCR-engineered PBMC when administered with nivolumab home and expand in secondary lymphoid organs and tumor deposits.

III. Clinical antitumor activity recording objective response rate.

OUTLINE: This is a dose-escalation study of nivolumab.

CONDITIONING REGIMEN: Patients receive cyclophosphamide intravenously (IV) over 1 hour on days -5 to -4 and fludarabine phosphate IV over 15-30 minutes on days -4 to -1.

NY-ESO-1 TCR PBMC INFUSION: Patients receive NY-ESO-1 TCR PBMC IV on day 0.

NIVOLUMAB: Patients receive nivolumab IV over 60 minutes on day 0 or 1. Treatment repeats every 2 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity.

NY-ESO-1(157-165) PEPTIDE PULSED DENDRITIC CELL (DC): Patients receive NY-ESO-1(157-165) peptide pulsed DC intradermally (ID) on days 1, 14, and 28.

LOW DOSE ALDESLEUKIN ADMINISTRATION: Patients receive aldesleukin subcutaneously (SC) twice daily (BID) for 7 days beginning on day 1 for a maximum of 14 doses.

After completion of study treatment, patients are followed up at least every 6 months for 3 years and then at least every 12 months for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Stage IV or locally advanced histologically confirmed solid tumors for which no alternative therapies with proven survival advantage are available
* At least 1 lesion amenable for outpatient biopsies; this should be a cutaneous or palpable metastatic site or a deeper site accessible by image-guided biopsy that is deemed safe to access by the treating physicians and interventional radiologists; patients without accessible lesions for biopsy but with prior tissue available from metastatic disease would be eligible at the investigator's discretion
* NY-ESO-1 positive malignancy by immunohistochemistry (IHC) utilizing commonly available NY-ESO-1 antibodies
* Human leukocyte antigen (HLA)-A*0201 (HLA-A2.1) positivity by molecular subtyping
* Age greater than or equal to 16 years old
* A minimum of one measurable lesion defined as:

  * Meeting the criteria for measurable disease according to Response Evaluation Criteria In Solid Tumors (RECIST)
  * Skin lesion(s) selected as non-completely biopsied target lesion(s) that can be accurately measured and recorded by color photography with a ruler to document the size of the target lesion(s)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Absolute neutrophil count >= 1.5 x 10^9 cells/L
* Platelets >= 100 x 10^9/L
* Hemoglobin >= 9 g/dL
* Aspartate and alanine aminotransferases (AST, ALT) =< 2.5 x upper limit of normal (ULN) (=< 5 x ULN, if documented liver metastases are present)
* Total bilirubin =< 2 x ULN (except patients with documented Gilbert's syndrome)
* Creatinine < 2 mg/dl (or a glomerular filtration rate > 60)
* Must be willing and able to accept two leukapheresis procedures
* Must be willing and able to provide written informed consent

Exclusion Criteria:

* Previously known hypersensitivity to any of the agents used in this study
* Received systemic treatment for cancer, including immunotherapy, within one month prior to initiation of dosing within this protocol
* History of, or significant evidence of risk for, chronic inflammatory or autoimmune disease (eg, Addison's disease, multiple sclerosis, Graves disease, Hashimoto's thyroiditis, inflammatory bowel disease, psoriasis, rheumatoid arthritis, systemic lupus erythematosus, hypophysitis, pituitary disorders, etc.); patients will be eligible if prior autoimmune disease is not deemed to be active (e.x. fibrotic damage of the thyroid after thyroiditis or its treatment, with stable thyroid hormone replacement therapy); vitiligo will not be a basis for exclusion
* History of inflammatory bowel disease, celiac disease, or other chronic gastrointestinal conditions associated with diarrhea or bleeding, or current acute colitis of any origin
* Potential requirement for systemic corticosteroids or concurrent immunosuppressive drugs based on prior history or received systemic steroids within the last 2 weeks prior to enrollment (inhaled or topical steroids at standard doses are allowed)
* Human immunodeficiency virus (HIV) seropositivity or other congenital or acquired immune deficiency state; if there is a positive result in the infectious disease testing that was not previously known, the patient will be referred to their primary physician and/or infectious disease specialist
* Hepatitis B or C seropositivity with evidence of ongoing liver damage; if there is a positive result in the infectious disease testing that was not previously known, the patient will be referred to their primary physician and/or infectious disease specialist
* Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol
* Known clinically active brain metastases; prior evidence of brain metastasis successfully treated with surgery or radiation therapy will not be exclusion for participation as long as they are deemed under control at the time of study enrollment and there are no neurological signs of potential brain metastases
* Pregnancy or breast-feeding; female patients must be surgically sterile or be postmenopausal for two years, or must agree to use effective contraception during the period of treatment and 6 months after; all female patients with reproductive potential must have a negative pregnancy test (serum/urine) within 24 hours from starting the conditioning chemotherapy; the definition of effective contraception will be based on the judgment of the study investigators; patients who are breastfeeding are not allowed on study
* Since IL-2 is administered following cell infusion:

  * Patients will be excluded if they have a history of clinically significant electrocardiogram (ECG) abnormalities, symptoms of cardiac ischemia or arrhythmias and have a left ventricular ejection fraction (LVEF) < 45% on a cardiac stress test (stress thallium, stress multi gated acquisition scan [MUGA], dobutamine echocardiogram, or other stress test)
  * Similarly, patients who are >= 50 years old with a baseline LVEF < 45% will be excluded
  * Patients with ECG results of any conduction delays (PR interval > 200 ms, corrected QT interval [QTC] > 480 ms), sinus bradycardia (resting heart rate < 50 beats per minute), sinus tachycardia (heart rate > 120 beats per minute) will be evaluated by a cardiologist prior to starting the trial; patients with any arrhythmias, including atrial fibrillation/atrial flutter, excessive ectopy (defined as > 20 premature ventricular contractions [PVCs] per minute), ventricular tachycardia, third (3rd) degree heart block will be excluded from the study unless cleared by a cardiologist
  * Patients with pulmonary function test abnormalities as evidenced by a forced expiration volume in one second (FEV1)/forced vital capacity (FVC) < 70% of predicted for normality will be excluded
* Evidence of diverticulitis at baseline, including evidence limited to computed tomography (CT) scan only
* Received 3 or more prior myelotoxic treatment regimens
* Bone marrow involvement based on CT or PET scan at screening

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2019-04-08 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events, defined following the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 15 years
  Simple descriptive statistics will be used to summarize toxicities observed after TCR transgenic cell infusion in terms of type (organ affected or laboratory determination such as absolute neutrophil count), severity and nadir or maximum values for the laboratory measures, time of onset (i.e. course number), duration, and reversibility or outcome. Tables will be created to summarize these toxicities and side effects by dose and by course.
Maximum tolerated dose based on dose-limiting toxicity using the Common Toxicity Criteria | First 60 days after ACT

SECONDARY OUTCOMES:
Feasibility of generating NY-ESO-1 TCR cells and/or NY-ESO 1(157-165) peptide pulsed DC vaccine, determined by the incidence of preparation not meeting the lot release criteria | 1 month
  Descriptive statistics including simple summary measures and plots appropriate for longitudinal data will be used.
Transgenic cell persistence | Up to 15 years
  Analysis will be performed both using immune monitoring and molecular techniques. Detection of surface expression of the NY-ESO-1 TCR transgenic protein will be analyzed both by major histocompatibility complex tetramer or dextramer analysis and staining for the specific region. Molecular analysis of the persistence of cells bearing the NY-ESO-1 TCR complementary deoxyribonucleic acid will be done by real time polymerase chain reaction techniques using primers specific for the transgenes and retroviral vector sequences. This testing will provide data to estimate the in vivo survival of lymphoc

OTHER OUTCOMES:
Antitumor activity as determined by RECIST | Up to 15 years
  The rate of complete response (CR) plus partial response (PR) will be used to explore antitumor activity. Response assessment will be performed by comparing standard CT imaging scans and photographs of target lesions from baseline with repeated imaging tests obtained by day +56 (8 weeks) after the TCR transgenic PBMC adoptive transfer, and then approximately every 2-3 months thereafter. To account for the frequently observed delayed responses with immunotherapy, patients with transient disease stabilization or progression by day 56 who do not receive further therapy but go on to meet RECIST cr
NY-ESO-1 TCR transgenic cell tumor trafficking (imaging) using 18F-FDG PET | Up to 40 days
  Regional uptake of 18F-FDG within metastatic tumor sites and secondary lymphoid organs will be quantified by standard uptake value (SUV) normalized to the body weight of the patient. As an internal quality control, SUVs will also be determined for several normal organs, such as muscle, liver and lungs. Findings with non-invasive molecular imaging will be compared with results from immune monitoring assays in blood samples and tumor biopsies at different intervals after NY-ESO-1 TCR ACT.

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Ribas, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frankiw L, Singh A, Peters C, Comin-Anduix B, Berent-Maoz B, Macabali M, Shammaie K, Quiros C, Kaplan-Lefko P, Baselga Carretero I, Ribas A, Nowicki TS. Immunotherapy resistance driven by loss of NY-ESO-1 expression in response to transgenic adoptive cellular therapy with PD-1 blockade. J Immunother Cancer. 2023 May;11(5):e006930. doi: 10.1136/jitc-2023-006930. PMID 37156551